CLINICAL TRIAL: NCT05404802
Title: Therapeutic Effectiveness of PARO Companion Robot for Elderly With Mild Cognitive Impairment/Dementia in Elderly Residential Setting: A Quasi-experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HKU_robot_protocol_v3
Record Dates: First submitted 2022-05-26; First posted 2022-06-03 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Technology
Keywords: Gerontechnology; Smart Healthcare Device; Digital Health Technology

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to the experimental group or the control group according to their floor of the residential care homes. The participants in the experimental group will be arranged to join the PARO intervention in Week 1 to 10. The control group will be arranged to attend 2 PARO training sessions after all assessments are completed.
Who Masked: Outcomes Assessor
Masking Description: Participants, training session moderators and observers of PARO sessions cannot and will not be blinded to the intervention. Assessors of the follow-up outcomes and the research analysts will not be involved in the recruitment and intervention delivery and will be blinded to the group allocation (single blindness).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Training sessions
  Each training session will last for 30-45 minutes, twice a week over a 10-week period in Week 1 to Week 10. Each session will be attended by a cluster of 4 to 6 participants, and each participant will have one PARO.
  Free-play sessions
  Two 15-30 minutes free-play sessions in each week of the 10 weeks are conducted on days when there are no training sessions.
  Interventions: Device: Experimental group intervention
- Control Group (Experimental): Training sessions
  Each training session will last for 30-45 minutes, once a week over a 2-week period after all assessments are completed. Each session will be attended by a cluster of 4 to 6 participants, and each participant will have one PARO.
  There is no free-play sessions for control group.
  Interventions: Device: Control group intervention

INTERVENTIONS:
Device: Experimental group intervention — Training session
  Facilitators will facilitate participants' interaction with PARO for 7 main activities, namely: (1) hugging PARO; (2) expressing emotions to PARO: (3) remembering PARO; (4) feeding PARO; (5) sleeping PARO; (6) bathing PARO; (7) decorating PARO.
  Free-play session
  In these sessions, every participant can interact with one PARO without instructions but are under the safety supervision of a PARO facilitator.
  Arms: Experimental Group
Device: Control group intervention — Facilitators will facilitate participants' interaction with PARO for 7 main activities, namely: (1) hugging PARO; (2) expressing emotions to PARO: (3) remembering PARO; (4) feeding PARO; (5) sleeping PARO; (6) bathing PARO; (7) decorating PARO.
  Arms: Control Group

SUMMARY:
The main trial is a 2-group quasi-experimental trial of comparing the outcome indicators between joining and not joining the 10-week personal assistive robot (PARO) training program in residents with dementia or mild cognitive impairment (MCI). The study questions are as follows:

Primary study questions:

i. Can participation of the 10-week PARO training program reduce neuropsychiatric symptoms at week 10?

ii. Can participation of the 10-week PARO training program reduce loneliness at week 10?

Secondary study questions:

iii. Can participation of PARO training session reduce pulse rate (as an indicator of stress and anxiety)?

iv. Can participation of PARO training session improve oxygen saturation (as an indicator of stress and anxiety)?

v. What are the participants' emotions and engagement in PARO training sessions?

Auxiliary study questions:

vi. Can participation of the 10-week PARO training program reduce neuropsychiatric symptoms at week 14?

vii. Can participation of the 10-week PARO training program reduce loneliness at week 14?

viii. Can participation of the 10-week PARO training program improve quality of life at week 10?

ix. Can participation of the 10-week PARO training program improve quality of life at week 14?

x. Can participation of the 10-week PARO training program improve sleep quality at week 10?

xi. Can participation of the 10-week PARO training program improve sleep quality at week 14?

xii. Can participation of the 10-week PARO training program improve cognitive functioning at week 10?

xiii. Can participation of the 10-week PARO training program improve cognitive functioning at week 14?

xiv. What are the feelings, satisfaction, and acceptance of PARO of the participants and PARO facilitators?

DETAILED DESCRIPTION:
Study design

This is a 2-group quasi-experimental trial of comparing the outcome indicators between joining and not joining the 10-week PARO training program in residents with dementia or mild cognitive impairment (MCI) in Haven of Hope Woo Ping Care & Attention Home. Residents from the Haven of Hope Hang Hau Care and Attention Home for Severely Disabled will also be recruited and join the PARO training program, but their data will be analysed independently. The feelings, satisfaction, and acceptance of PARO of the participants and PARO facilitators.

Procedures

Training of PARO facilitators

Nurses, social workers, occupational therapists, health care assistants and program workers of the service units will be recruited and trained as PARO facilitators. The formal PARO facilitator training lasts for about 3 hours. An intervention protocol will be provided for the facilitators in running the training sessions.

Participants' recruitment and consent

In the residential care homes under Haven of Hope Christian Service (HOHCS), the care staff and nurses will check the eligibility of the elderly and invite eligible participants to join the trial. Residents scoring above the cutoff for dementia in Montreal Cognitive Assessment (MoCA) and not receiving a medical diagnosis of dementia or other mentally incapacitating disease will be classified as competent in giving consent. For residents scoring below the cutoff in MoCA or receiving a diagnosis of mentally incapacitating disease, we will follow the criteria stated in the Alzheimer Europe Report (2011) to ensure that they are provided chances to give consent. In particular, four criteria will be evaluated, including 1) the person must have sufficient capacity to understand the information, 2) the person is able to retain, use and weight up such information for making a decision, 3) the person will understand the benefit, risk, and convenience, 4) the person must have the ability to communicate the decision. The University of Hong Kong (HKU) research staff and the care staff will first commit them in a causal chat to assess their ability to communicate and understand the dialogues.

If residents are competent in giving consent, both residents and their family members, will be approached for consent. In cases residents are not competent in giving consents, only their family members will be approached for consent. They will then be referred to join a 1-to-1 study introduction session. In this session, HKU research staff and service unit staff will introduce the study to the participant, and invite them to sign a consent form.

After the consent is obtained, the HKU research staff will assist the participant to complete the UCLA 3-Item Loneliness Scale (UCLA 3-item), Mini-Mental State Examination (MMSE), the 5-level EQ-5D version (EQ-5D-5L), and Insomnia Severity Index (ISI), and assist the care staff to complete Neuropsychiatric Inventory Questionnaire (NPI-Q). Participants will be allocated to the experimental group or the control group according to their floor of the residential care homes. The participants in the experimental group will be arranged to join the PARO intervention in Week 1 to 10. The control group will be arranged to attend 2 PARO training sessions after all assessments are completed. As a voluntary participation, the participants have the right to withdraw from the study and intervention any time without consequences.

Interventions

Training sessions for experimental group

Each session aims to facilitate engagement, communication and interaction with the robots and other participants. Each session will take place for 30-45 minutes, twice a week over a 10-week period. Each session will be attended by a cluster of 4 to 6 participants. In each session, several activities with PARO will be supervised by the facilitator including baby-sitting PARO, feeding PARO, grooming PARO, etc. The first session will be used as a pilot run to revise our test protocol. The first three group sessions will be primarily focused on enhancing the intimacy between the group participants and their therapeutic relationship with the PARO companion robot. Participants will be introduced with the PARO training program and each other, followed by naming PARO. Fun activities such as informing each other of one's Chinese zodiac and animal's name matching game will be used to develop their friendliness and rapport towards PARO. In the third session, the facilitators will show seal photos and videos (*subject to the availability of audio-visual (AV) equipment in the care homes) so that participants will be able to recognise PARO.

Facilitators will facilitate participants' interaction with PARO for 7 main activities, namely: (1) hugging PARO: (1a) touching and hugging PARO; (1b) comparing PARO with a pet; (2) expressing emotions to PARO: (2a) selecting seven emotional stickers and talking about emotions; (2b) observing positive/negative reactions of PARO; (3) remembering PARO: (3a) talking about PARO's name and seal; (3b) becoming accustomed to PARO's movements, noises, etc; (4) feeding PARO: (4a) searching animal's feed, (4b) sharing food and snacks, (4c) feeding PARO; (5) sleeping PARO: (5a) sing favourite song or singing and clapping song, (5b) putting PARO to sleep with a cradle song; (6) bathing PARO: (6a) cleaning hands, (6b) cleaning PARO, (6c) combing PARO's hair; (7) decorating PARO: (7a) decorating PARO with ribbon, scarf, cap, etc., (7b) decorating oneself with favourite things.

Free-play sessions

For the experimental group, during the 10-week training program, to increase the exposure of participants in experimental group to PARO, two 15-30 minutes free-play sessions in each week are conducted on days when there are no training sessions. In these sessions, every participant can interact with one PARO without instructions but are under the safety supervision of a PARO facilitator.

Intervention for control group

Control group will receive no PARO-related intervention from week 1 to week 10. They will attend 2 training sessions after all assessments are completed. Activity content in these training sessions will be similar to those for the experimental group.

Data collection

HKU research staff who are blinded to the group allocation will administer all the questionnaires at baseline, 10-week and 14-week. For experimental group, after each training session and free-play session, PARO facilitators will complete Engagement of a Person with Dementia Scale (EPDS) for every participant. After each training session, they will complete two items about compliance and non-compliance with instructions for every participant. There were three selected training sessions in every cluster in the beginning phase, middle phase and ending phase that biomarkers will be collected and process observed by HKU senior research assistant. The biomarkers of pulse rate and oxygen saturation of the participants (as an indicator of feelings of stress and anxiety) will be measured using pulse oximeter before and after each of the three selected training sessions. The emotions of every participant and any special events during the three selected training sessions will be documented by HKU senior research assistant using Observed Emotion Rating Scale (OERS). To reduce the possible impacts brought by the presence of research team, the observer will introduce himself before and after the residents move to the activity room. Also, the observer will not interfere into the training activities.

In case of events (e.g. COVID-19) that prohibit HKU research staff to conduct assessment on site, assessment will be conducted via online communication apps (e.g. Zoom), and processes of training sessions will be video-recorded,

Qualitative interview

To collect feedback towards the PARO companion robot intervention, we will use purposive sampling to select 10 participants and at most 6 facilitators to conduct semi-structured qualitative interviews to collect opinion on their satisfaction and perceived acceptance on PARO features. An interview guide with open-ended and iterative questions will be used to probe for more experiences from the interviewees. Each interview will be conducted by a trained research assistant and will last about 30 minutes.

Blinding

Participants, training session moderators and observers of PARO sessions cannot and will not be blinded to the intervention. Assessors of the follow-up outcomes and the research analysts will not be involved in the recruitment and intervention delivery and will be blinded to the group allocation (single blindness).

Sample size determination

The sample size is estimated by the current number of dementia/MCI residents in the test sites. In the Woo Ping Care & Attention Home, 52 residents have been diagnosed dementia/MCI. In the Care and Attention Home for Severely Disabled, 5 have been diagnosed. Therefore, the study will include 57 residents in total.

Data analyses

Main analysis

Linear mixed model analysis will be used to test the interaction between group and time. A partial-eta square will be used to estimate the effect size of the outcome indicators in comparing the intervention group with the control group.

Process evaluations

For the biomarkers, linear mixed model analysis will be used to test the interaction between group and time. A partial-eta square will be used to estimate the effect size of the outcome indicators in comparing the intervention group with the control group. For the rated scales, descriptive statistics will be used to show the changes of emotions and incidence of negative emotions.

Qualitative interview

The interview content will be transcribed verbatim in Chinese for further analysis. We will analyze the qualitative interview transcripts using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of the PARO training program. The results will then be discussed and consolidated in the panel meetings with the co-authors.

ELIGIBILITY:
Inclusion Criteria for residents in main trial:

* Is diagnosed with mild to moderate dementia by doctors
* Score at least 5 (Pan et al., 2020) and lower than the norm-derived age and education adjusted cutoff scores 7th percentile in HK-MoCA (Wong et al., 2015), non-dementia patients

Exclusion Criteria for residents in main trial:

* Have unstable physical or psychological conditions as advised by doctors or nurse in charge
* Have severe medical conditions which limit the ability to participate in the PARO sessions
* Have visual or hearing impairment that interfere with cognitive intervention
* Fear or reluctance in using robots
* Unable to communicate

Inclusion Criteria for residents in qualitative interviews:

* Have participated in the main trial
* Able to verbally communicate in Cantonese as perceived by the staff of the related home

Exclusion Criteria for residents in qualitative interviews:

* None

Inclusion Criteria of PARO facilitator for qualitative interviews:

* Have participated in the main trial

Exclusion Criteria for PARO facilitator in qualitative interviews:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
10 week change in neuropsychiatric symptoms after participating in 10-week PARO training program | Baseline and the 10th week
  Change of neuropsychiatric symptoms after participating in 10-week PARO training program will be measured by Neuropsychiatric Inventory Questionnaire (NPI-Q; Cummings, et al., 1994; Kauffer, 1999). The range of the the severity scale is 12 to 36, with higher score indicating more severe neuropsychiatric symptoms. The range of the caregiver distress scale is 0 to 60, with higher score indicating higher caregiver distress.
10 week change in loneliness after participating in 10-week PARO training program | Baseline and the 10th week
  Change of loneliness after participating in 10-week PARO training program will be measured by UCLA Loneliness Scale 3 items (UCLA 3-items, Russell et al., 1980; Liu et al., 2020). The minimum and maximum values of the scale are 3 and 9 respectively, with higher score indicating higher level of loneliness.

SECONDARY OUTCOMES:
Change in feelings of stress and anxiety as indicated by pulse rate after participating in PARO training session | Before and after the three training sessions during the 10-week trial period
  The change of feelings of stress and anxiety after participating in PARO training session will be measured by pulse rate.
Change in feelings of stress and anxiety as indicated by oxygen saturation after participating in PARO training session | Before and after the three training sessions during the 10-week trial period
  The change of feelings of stress and anxiety after participating in PARO training session will be measured by oxygen saturation
Qualitative Measure: Observed emotions | 3 PARO training sessions during the 10-week trial period
  Emotions will serve as an indicator of satisfaction and acceptance of PARO, and will be observed in PARO training session using Observed Emotion Rating Scale (OERS; Lawton et al., 1999). Under the scale, the 5 emotions of pleasure, general alertness, anxiety/ fear, anger, and sadness are observed. The minimum and maximum values of each coding for 10 minutes observation are 1 and 5 respectively, with higher score indicating longer duration of the observed emotion within the 10 minute period.
Qualitative Measure: Observed engagement | Every PARO training session and every free-play session during the 10-week trial period
  Engagement will serve as an indicator of satisfaction and acceptance of PARO. After each training session and free-play session, PARO facilitators will complete Engagement of a Person with Dementia Scale (EPDS; Jones et al., 2018) for every participant. The minimum and maximum values of EPDS are 10 and 50 respectively, with higher score indicating higher level of positive engagement exhibited.
Qualitative Measure: Observed engagement (compliance) | Every PARO training session during the 10-week trial period
  Compliance will serve as an indicator of engagement, satisfaction and acceptance of PARO. After each training session and free-play session, PARO facilitators will complete two items about compliance and non-compliance with instructions for every participant. The minimum and maximum values of the sum of the two items are 2 and 10 respectively, with higher score indicating higher compliance.
14 week change in neuropsychiatric symptoms after participating in 10-week PARO training program | Baseline and 14th week
  Change of neuropsychiatric symptoms after participating in 10-week PARO training program will be measured by Neuropsychiatric Inventory Questionnaire (NPI-Q; Cummings, et al., 1994; Kauffer, 1999). The range of the the severity scale is 12 to 36, with higher score indicating more severe neuropsychiatric symptoms. The range of the caregiver distress scale is 0 to 60, with higher score indicating higher caregiver distress.
14 week change in loneliness after participating in 10-week PARO training program | Baseline and 14th week
  Change of loneliness after participating in 10-week PARO training program will be measured by UCLA Loneliness Scale 3 items (UCLA 3-items, Russell et al., 1980; Liu et al., 2020). The minimum and maximum values of the scale are 3 and 9 respectively, with higher score indicating higher level of loneliness.
Change in quality of life after participating in 10-week PARO training program | Baseline, the 10th week and 14th week
  The change of quality of life after participating in 10-week PARO training program will be measured by 5-level EQ-5D (EQ-5D-5L; Wong et al., 2018). Using the algorithm based on Hong Kong population, the minimum and maximum utility values of the scale are -0.803 and 1 respectively, with higher score indicating better quality of life.
Change in sleep quality after participating in 10-week PARO training program | Baseline, the 10th week and 14th week
  The change of sleep quality after participating in 10-week PARO training program will be measured by Insomnia Severity Index (ISI; Morin 1993; Yu, 2010). The minimum and maximum values of the scale are 0 and 16 respectively, with higher score indicating higher insomnia severity.
Change in cognitive functions after participating in 10-week PARO training program | Baseline, the 10th week and 14th week
  The change of cognitive functions of after participating in 10-week PARO training program will be measured by Mini-Mental State Examination (MMSE; Folstein et al., 1975). The minimum and maximum values of the scale are 0 and 30 respectively, with higher score indicating higher level of cognitive functioning.
Qualitative Measure: Perceived feelings, satisfaction and acceptance on companion robot by the participants | within 2 weeks after week 10
  The participants answer the following question in semi-structured qualitative interviews:
  1. Do you like (the name of the robot)?
  2. What do you like about (the name of the robot)?
  3. Did (the name of the robot) do something you dislike?
  4. Is there anything you dislike about (the name of the robot)?
  5. How do you feel with the company of (the name of the robot)?
  6. What do you do with (the name of the robot) regularly?
  7. Do you wish to spend more time (the name of the robot)?
  8. Under what circumstances, do you need the company of (the name of the robot)
  9. Do you wish or need others to spend time with (the name of the robot) and you?
  10. To conclude, are you satisfied or dissatisfied with (the name of the robot)?
  11. Do you wish to see it again?
Qualitative Measure: Perceived feelings, satisfaction and acceptance on companion robot by the PARO facilitators | within 2 weeks after week 10
  The PARO facilitators answer the following questions in semi-structured qualitative interviews:
  1. Were the companion robots safe?
  2. Was it easy or difficult to use the companion robots?
  3. Did you expect the participants to accept the companion robots?
  4. What types of participants are more likely and less likely to accept the companion robots?
  5. When are the participants more willing to interact with the companion robots?
  6. What do you suggest to improve the acceptability of the companion robots?
  7. Is the training on companion robots sufficient?
  8. What did you expect to be the benefits and concerns of the companion robots?
  9. Did you find these benefits and concerns?
  10. Were there any unexpected benefits and concerns?
  11. What are your suggestions to the staff who will use the companion robots?
  12. Are you satisfied or dissatisfied with the companion robots?
  13. Do you want to use the companion robots in the future?
  14. Are companion robots cost-effective?

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Haven of Hope Hang Hau Care and Attention Home for Severely Disabled, Hong Kong
  - Haven of Hope Woo Ping Care & Attention Home, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.

REFERENCES:
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Jones C, Sung B, Moyle W. Engagement of a Person with Dementia Scale: Establishing content validity and psychometric properties. J Adv Nurs. 2018 May 17. doi: 10.1111/jan.13717. Online ahead of print. PMID 29772602
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] Lawton MP, Van Haitsma K, Klapper J. Observed affect in nursing home residents with Alzheimer's disease. J Gerontol B Psychol Sci Soc Sci. 1996 Jan;51(1):P3-14. doi: 10.1093/geronb/51b.1.p3. PMID 8548515
- [Background] Pan IMY, Lau MS, Mak SC, Hariman KW, Hon SKH, Ching WK, Cheng KM, Chan CF. Staging of Dementia Severity With the Hong Kong Version of the Montreal Cognitive Assessment (HK-MoCA)'s. Alzheimer Dis Assoc Disord. 2020 Oct-Dec;34(4):333-338. doi: 10.1097/WAD.0000000000000399. PMID 32701514
- [Background] Piau A, Campo E, Rumeau P, Vellas B, Nourhashemi F. Aging society and gerontechnology: a solution for an independent living? J Nutr Health Aging. 2014 Jan;18(1):97-112. doi: 10.1007/s12603-013-0356-5. PMID 24402399
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Wong A, Law LS, Liu W, Wang Z, Lo ES, Lau A, Wong LK, Mok VC. Montreal Cognitive Assessment: One Cutoff Never Fits All. Stroke. 2015 Dec;46(12):3547-50. doi: 10.1161/STROKEAHA.115.011226. Epub 2015 Oct 15. PMID 26470772
- [Background] Carmeli E. Aspects of assistive gerontechnology. Int J Disabil Hum Dev. 2009; 8(3): 215-218.
- [Background] Liu T, Lu S, Leung DKY, Sze LCY, Kwok WW, Tang JYM, Luo H, Lum TYS, Wong GHY. Adapting the UCLA 3-item loneliness scale for community-based depressive symptoms screening interview among older Chinese: a cross-sectional study. BMJ Open. 2020 Dec 10;10(12):e041921. doi: 10.1136/bmjopen-2020-041921. PMID 33303463
- [Background] Yu DS. Insomnia Severity Index: psychometric properties with Chinese community-dwelling older people. J Adv Nurs. 2010 Oct;66(10):2350-9. doi: 10.1111/j.1365-2648.2010.05394.x. Epub 2010 Aug 16. PMID 20722803
- [Background] Morin CM. Insomnia: psychological assessment and management. Guilford press. 1993.
- [Background] Wong ELY, Ramos-Goni JM, Cheung AWL, Wong AYK, Rivero-Arias O. Assessing the Use of a Feedback Module to Model EQ-5D-5L Health States Values in Hong Kong. Patient. 2018 Apr;11(2):235-247. doi: 10.1007/s40271-017-0278-0. PMID 29019161